CLINICAL TRIAL: NCT06467487
Title: Leveraging Community Engagement and Electronic Health Record Strategies to Promote Diverse Participation in COVID-19 Clinical Trials -2
Brief Title: Electronic Health Record Strategies to Promote Diverse Participation in Research AIM 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000032716_a; 75F40120C00174 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Patient Participation
Keywords: Online Patient Portal
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Optimized Letter (Experimental): Participants receive an 'optimized' letter.
  Interventions: Other: Optimized Letter
- Optimized Message (Experimental): Participants receive an 'optimized' message.
  Interventions: Other: Direct to Patient Message - Optimized
- Optimized Letter + Optimized Message (Experimental): Participants receive both a 'optimized' letter and a 'optimized' message.
  Interventions: Other: Optimized Letter; Other: Direct to Patient Message - Optimized
- Generic Letter (Active Comparator): Participants receive a 'usual' letter.
  Interventions: Other: Traditional Letter
- Generic Message (Active Comparator): Participants receive a 'usual' message.
  Interventions: Other: Direct to Patient Message
- Generic Letter + Generic Message (Experimental): Participants receive both a 'usual' letter and a 'usual' message.
  Interventions: Other: Traditional Letter; Other: Direct to Patient Message

INTERVENTIONS:
Other: Traditional Letter — Patients receive a traditional letter.
  Arms: Generic Letter; Generic Letter + Generic Message
Other: Direct to Patient Message — Patients receive a direct to patient message via the portal.
  Arms: Generic Letter + Generic Message; Generic Message
Other: Optimized Letter — Patients receive an optimized letter.
  Arms: Optimized Letter; Optimized Letter + Optimized Message
Other: Direct to Patient Message - Optimized — Patients receive an optimized direct to patient message via the portal.
  Arms: Optimized Letter + Optimized Message; Optimized Message

SUMMARY:
Based on the outcomes of the initial study (NCT05348603), this optimization study will employ the most effective interventions (letters and messages) and distribute these communications to underrepresented minorities to further promote interest in research. Optimized language will be distributed in English, Spanish, Portuguese, Chinese, Arabic, or Haitian Creole, based on preferred language identified in the patient profile in an electronic medical records system.

DETAILED DESCRIPTION:
The primary objective of the optimization study is to examine the effectiveness on increasing interest in research of an optimized letter versus a generic letter; an optimized message versus a generic message; and an optimized letter and an optimized message versus a generic letter and a generic message.

The secondary objective of the optimization study is to examine the effectiveness on increasing participation in research of an optimized letter versus a generic letter, an optimized message versus a generic message, an optimized letter and an optimized message versus a generic letter and a generic message.

ELIGIBILITY:
Inclusion Criteria:

* Has an account with the online patient portal
* Has logged into the online patient portal at least once in the past year
* Has not set up a research profile

Exclusion Criteria:

* Currently enrolled in a clinical trial
* Opted out of research
* On active cancer treatment
* Active member of the study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214526 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Number of patients who create a research profile | 12 months
  The outcome will be assessed by querying the patient's electronic medical record to determine whether the patient has registered in the Yale University Volunteer Database. This database is comprised of patients who agree to be contacted if there is a study at Yale that meets their interests.

SECONDARY OUTCOMES:
Number of patients who enroll in a research study | 12 months
  The outcome will be assessed by querying our clinical trials management system or electronic health record system to determine if the patient has consented to participate in a research study.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Smith, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No